CLINICAL TRIAL: NCT06116487
Title: Evaluation of Magnetic Resonance Imaging as Alternative to Cone Beam Computed Tomography for the Assessment of Furcation Involvement in Molars
Brief Title: MRI as Alternative to CBCT for the Assessment of Furcation Involvement in Molars
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Elias Salzmann, Principal Investigator, Medical University of Vienna
Other Study IDs: 1208/2023
Record Dates: First submitted 2023-10-25; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis; Periodontal Diseases; Furcation Defects
Keywords: CBCT; MRI; Furcation involvement
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Furcation Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of this prospective study is to compare magnetic resonance imaging (MRI) and cone beam computed tomography (CBCT) to diagnose furcation involvement (FI) in molars in patients with periodontitis. The focus is on the differentiation of grad II and III according to Hamp et al. 1975. 140 molars (70 upper and 70 lower) will be investigated with CBCT and MRI. Due to the absence of ionic radiation MRI might be a radiation free diagnostic tool to assess FI in the future without harmful radiation for the patient. Patients of the Dental Clinic, Medical University of Vienna, who need a CBCT and have a clinically diagnosed FI can be a participant of this clinical trial and do in addition to their CBCT a MRI. The accuracy of MRI will be compared to the diagnostic gold standard CBCT. If patients need additional periodontal treatment, e.g., periodontal surgery, a subgroup will also be analysed with intraoperative measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FI grade II or III, patients who need a CBCT, not pregnant

Exclusion Criteria:

* Patients with contraindications to perform a MRI

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with clinical detected furcation involvement at the first or second molars
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
horizontal furcation defects according to Hamp 1975 | day 1
  Grad 0, I, II, III

SECONDARY OUTCOMES:
horizontal bone loss | day 1
  measured in mm
vertical bone loss | day 1
  measured in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Clinic of Dentistry, Vienna, Austria